CLINICAL TRIAL: NCT03630406
Title: Vaginal Elasticity Assessment Before and After Vaginal Carbon Dioxide Laser Treatment.as Measured by Vaginal Tactile Imaging.
Brief Title: Vaginal Elasticity Assessment Before and After Vaginal Carbon Dioxide Laser Treatment.
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Primary Investigator, Rambam Health Care Campus
Other Study IDs: 0022-18-RMB
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Laser Burn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laser treatment: Female patients with either SUI of vaginal wall weakness and prolapse refered for an attempt at laser treatment.
  Interventions: Diagnostic Test: Vaginal Tactile Imaging

INTERVENTIONS:
Diagnostic Test: Vaginal Tactile Imaging — Vaginal Tactile Imaging

SUMMARY:
Female patients with either stress urinary incontinence (SUI) or vaginal wall weakness and prolapse will be evaluated for vaginal elasticity using vaginal tactile imaging both before and after Carbon Dioxide laser treatment.

DETAILED DESCRIPTION:
Patients will be recruited and sign a consent form. The patients included are patients with SUI or vaginal wall weakness and prolapse. Each participant undergoes 3 laser treatments 4 weeks apart.

Assessment of vaginal elasticity via vaginal tactile imaging will be performed at 3 different points:

* Before the first treatment session (baseline).
* Before and after each treatment session.
* 3 months post final treatment. Every patient will serve as her own control. Demographic, gynecologic and obstetric history will be obtained from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Any woman undergoing vaginal Carbon Dioxide laser treatment.

Exclusion Criteria:

* Women that are not in the age range.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients.
Study Population: Female patients with either SUI or vaginal wall weakness and prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Vaginal elasticity assessment | up to 3 months from enrollment
  Vaginal elasticity as measured by the vaginal tactile imager

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Principal Investigator
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided